CLINICAL TRIAL: NCT02008864
Title: Phase II Study of the Effect of Senna Alexandrina Mill. on Uremic Pruritus and Serum IL-2, INF-δ and TNF-α Levels of Hemodialysed Patients
Brief Title: Evaluating the Effect of Senna in Uremic Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pouya Faridi, Dr., Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Senna in Uremic Pruritus
Record Dates: First submitted 2013-12-01; First posted 2013-12-11 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: End Stage Renal Disease; Pruritus
Keywords: End stage renal diseases; Hemodialysis; Uremic pruritus; Iranian traditional medicine; Cassia angustifolia
MeSH Terms: conditions — Kidney Failure, Chronic; Pruritus | interventions — Sennosides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Wheat
  Interventions: Drug: Placebo
- Senna (Active Comparator): Senna
  Interventions: Drug: Senna

INTERVENTIONS:
Drug: Senna — (7.5 mg of sennosoides A and B) Senna tablet/ 2 times per day
  Arms: Senna
Drug: Placebo — Placebo tablet/ 2 times per day
  Arms: Placebo

SUMMARY:
Uremic pruritus remains one of the most frustrating and potentially disabling symptoms in patients with end stage renal disease. It affect up to 90 percent of patients with end stage renal disease. Several hypotheses have been postulated for the possible underlying etiology, but none is conclusive. Aside from kidney transplantation, which is only definitive treatment, therapeutic approaches have largely been empirical, and no firm evident-base treatments are available. The main goal of therapy remains to minimize severity of pruritus. In Iranian traditional medicine Cassia senna L. is used for healing uremic pruritus . In this study investigators considered to evaluate effect of Cassia senna L. in uremic pruritus by a double blind placebo control clinical trial. It is hypothesized that oral Cassia senna L. may attenuate uremic pruritus by decreasing serum IL-2, IFN-γ and TNF-α.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients
* Suffering from pruritus for at least 6 weeks
* Have not responded to other drugs

Exclusion Criteria:

* Dermatological disease
* Liver disease
* Metabolic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Severity of Pruritis, as measured by a visual analogue scale | 3 months
  A '0' score represented absence of pruritus and a '10' represented the greatest severity of symptoms.

SECONDARY OUTCOMES:
Serum IL-2 level | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jamshid Roozbeh, MD, Study Chair — Shiraz University of Medical Sciences; Abdolali Mohagheghzadeh, PhD, Principal Investigator — Shiraz University of Medical Sciences; Mohammad Mehdi Sagheb, MD, Principal Investigator — Shiraz University of Medical Sciences; Arian Kamali-Sarvestani, Pharm D, Study Director — Shiraz University of Medical Sciences; Pouya Faridi, PhD, Study Director — Shiraz University of Medical Sciences

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264